CLINICAL TRIAL: NCT00617812
Title: An Open Label Multicentric Study to Evaluate the Immunogenicity and Safety of Indigenously Developed DTPwHB-Hib (Liquid) Pentavalent Combination Vaccine (Shan 5) in Indian Infants.
Brief Title: Safety and Immunogenicity Study of a Liquid Pentavalent Combination Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shantha Biotechnics Limited (Industry)
Responsible Party: Head Clinical Research and Medical Affairs, Shantha Biotechnics Limited
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SBL/DTPwHB-Hib/PMS/2007/0100
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Haemophilus Influenzae Type B
Keywords: Vaccine; Prevention; Diphtheria; Tetanus; Pertussis; Hepatitis B; Haemophilus influenzae type b; Healthy infants
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Haemophilus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Shan5 (Experimental)
  Interventions: Biological: Shan5

INTERVENTIONS:
Biological: Shan5 — Diphtheria, tetanus, whole cell pertussis, recombinant hepatitis B and Hib tetanus toxoid conjugate pentavalent liquid combination vaccine

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of an indigenously developed liquid pentavalent (diphtheria, tetanus, pertussis, hepatitis B and Hib) combination vaccine in healthy Indian infants as a part of the routine immunization in accordance with the EPI schedule.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children in the age group six to eight weeks
* Born after a normal gestational period (36 - 42 weeks)
* Mother's HBsAg assured negative.
* Father, mother or legally acceptable representative properly informed about the study and having signed the informed consent form.
* Parents willing to fill the Diary Card

Exclusion Criteria:

* Administration of immunoglobulin or any blood products since birth.
* Use of any investigational, on-registered drug, or vaccine other than the study vaccine (with the exception of OPV & BCG vaccine) during the study period or within 30 days preceding the first dose of the study vaccine.
* Previous vaccination or evidence of infection with DTP.
* History of allergic disease or reaction likely to be exacerbated by any component of the vaccine including allergy to antibiotics.
* Major congenital or hereditary immunodeficiency.
* Infants having evidence of disease or fever, history of allergic disease or persistent hematological, hepatic, renal, cardiac or respiratory disease and signs of a CNS disorder at the time of vaccination.
* Infants showing any of the following reactions after any dose of study vaccine will be withdrawn for subsequent doses: body temperature more than 40.4 degree Celsius, persistent screaming or crying for 3 hours within 48 hours of vaccination, seizures, encephalopathy and hypersensitivity reaction.
* Parent/s or guardian of subject unable to maintain diary card
* Simultaneous participation in any other clinical study

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2008-03; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Seroprotection rates for Diphtheria, Tetanus, Pertussis, Hepatitis B and Hib following 3 doses of the vaccine. | 4 months

SECONDARY OUTCOMES:
Solicited and unsolicited local and systemic adverse events following vaccination | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Raman Rao, MD, Study Director — Shantha Biotechnics Limited, Hyderabad, India
Locations (4):
- India (4):
  - Deccan College of Medical Sciences, Hyderabaad, Andhra Pradesh
  - Ankur Institute of Child Health, Ahmedabad, Gujarat
  - JSS Medical College, Mysore, Karnataka
  - Institute of Child Health, Kolkata, West Bengal